CLINICAL TRIAL: NCT02248181
Title: Post Marketing Surveillance Study of Sifrol® - Monotherapy in Patients With Idiopathic Parkinson's Disease
Brief Title: Post Marketing Surveillance Study of Sifrol® in Patients With Idiopathic Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.539
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Idiopathic PD patients
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole
  Other Names: Sifrol®

SUMMARY:
Study to document pramipexole dosing during monotherapy, occurrence of fluctuations and dyskinesias, dose increases after deterioration of Parkinson's disease (PD) symptoms, assessment of the reasons for add-on treatment with L-Dopa and dosing of pramipexole and L-Dopa when given concomitantly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early stage idiopathic Parkinson's Disease
* No pre-treatment with any dopaminergic treatment (de novo patients), or Pre-treatment with L-Dopa at doses of < 200 mg/d

Exclusion Criteria:

* Treating physicians are asked to consider the regulation described in the Summary of Product Characteristics (SmPC) for the treatment with pramipexole

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Idiopathic PD patients recruited at office-based neurologists, psychiatrists or physicians in special neurological clinics
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2004-02; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in dosing details of Pramipexole | up to 21 months
Occurrence and clinical course of Parkinson Disease (PD) motor symptoms | up to 21 months

SECONDARY OUTCOMES:
Assessment of Kinetic Tremor | up to 21 months
  Spiral test with at least five rotations from the centre to the edge in blinded fashion
Change in dosing details of L-Dopa | up to 21 months
Global Assessment of tolerability by investigator on 4-point scale | after 21 months
Global assessment of efficacy by investigator on a 4-point scale | after 21 months
Number of patients with adverse drug reactions | up to 21 months